CLINICAL TRIAL: NCT03757819
Title: Can Transcranial Direct Stimulation Improve Walking in Multiple Sclerosis?
Brief Title: Transcranial Direct Current Stimulation and Walking in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thorsten Rudroff (Other)
Responsible Party: Sponsor-Investigator, Thorsten Rudroff, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 201810705
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Transcranial Direct Current Stimulation
Keywords: Multiple Scerosis
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This study employed a double-blind, sham-controlled, parallel-randomized crossover design. Each participant attended three sessions. In the first session, participants were consented and completed the Patient-Determined Disease State and Fatigue Severity Scale questionnaires. Then, after a counter-balanced randomization into BEFORE or DURING groups, the participants completed a 6-Minute Walk Test for baseline/familiarization purposes. The second and third sessions involved brain stimulation or sham stimulation either before or during a 6-Minute Walk Test, depending on group assignment. The brain stimulation was randomly assigned to either session two or three, and sham stimulation was performed in the other session.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Before Walking tDCS first then SHAM (Experimental): To investigate the effects of tDCS applied before walking versus during to evaluate effectiveness of the intervention.
  Interventions: Device: tDCS; Device: SHAM
- During Walking tDCS first then SHAM (Experimental): To investigate the effects of tDCS applied before walking versus during to evaluate effectiveness of the intervention.
  Interventions: Device: tDCS; Device: SHAM

INTERVENTIONS:
Device: tDCS — Brain Stimulation
Device: SHAM — Placebo device

SUMMARY:
Weakness on one side of the body is a hallmark of Multiple Sclerosis (MS), which has been determined to be a significant cause of progressive worsening of walking abilities. Currently, there are no efficient rehabilitation strategies available to target strength asymmetries and walking impairments. Many of the current treatments, including pharmaceuticals, are only mildly effective and are often very expensive. Thus, the development of practical, inexpensive, and effective adjunct treatments is needed.

The study is to examine the efficacy of different tDCS protocols at improving walking in PwMS. Although the details of the studies slightly vary, the global aspects of the experimental procedures are identical with the exception that the tDCS stimulation parameter timing differs between the groups. The study will be double-blind, sham-controlled, randomized cross-over design.

Maximal voluntary contractions (MVCs) of the right and left knee extensors, knee flexors, hip flexors, and dorsiflexors will be performed to determine the more-affected leg.

The study compromises 2 groups of subjects which will attend the lab for three sessions. In the first session subjects will be consented, complete the PDDS, the Fatigue Severity Scale (FSS), and a 6 minute walk test (6-MWT) for baseline performance. The second session will involve a 6 MWT performed in association with 2 conditions. Group 1: DURINGtDCS, DURINGSHAM. Group 2: BEFOREtDCS, BEFORESHAM. The conditions in each group will be in a randomized order. Intensity of tDCS will be 2mA for both groups. Group 1 will receive the conditions during the 6 MWT. tDCS for 6 min has been shown to be sufficient to induce cortical excitability. Group 2 will receive 13 min of tDCS or sham, which results in after effects lasting through the completion of the 6 MWT. tDCS will be applied to the motor cortex (M1) corresponding to the more-affected leg either before or during the 6 min walk test

DETAILED DESCRIPTION:
Prospective participants, men and women with MS, will be recruited. To accomplish this study, each of the two groups of participants will need to complete 3 sessions at the INPL, each separated by 5-8 days. The duration of each session will be approximately one hour. The investigators expect data collection to last 6 months.

The study compromises 2 groups of subjects which will attend the lab for three sessions. In the first session subjects will be consented, complete the Patient Determined Disease Steps (PDDS) questionnaire, the Fatigue Severity Scale (FSS), and a 6MWT for baseline performance. The second session will involve a 6 MWT performed in association with 2 conditions. Group 1: DURING_tDCS, DURING_SHAM. Group 2: BEFORE_tDCS, BEFORE_SHAM. tDCS will be applied first follwed by SHAM in each group. Intensity of tDCS will be 2mA for both groups. Group 1 will receive the conditions during the 6 MWT. tDCS for 6 min has been shown to be sufficient to induce cortical excitability. Group 2 will receive 13 min of tDCS or sham which results in after effects lasting through the completion of the 6MWT. tDCS will be applied to the motor cortex (M1)corresponding to the more-affected leg either before or during the 6 min walk test. Leg strength, 6 MWT, and tDCS: Maximal voluntary contractions (MVCs) of the right and left knee extensors, knee flexors, hip flexors, and dorsiflexors will be performed to determine the more-affected leg. When leg strength difference is less than 10%, the more affected side will be based on self-report. For the 6 MWT, participants will be asked to walk as far as they can in 6 minutes. The 6 MWT is well established in MS research and, in order to measure fatigability as a secondary outcome, the literature suggest using a 6MWT rather than a 2MWT.Participants will walk in a cordoned off hallway between two cones placed approximately 30 meters apart. The primary outcome measure will be the distance covered in the 6 MWT. Since the investigators hypothesize that tDCS will alter the utilization of their more-affected leg, standard gait metrics during the 6MWT including gait speed, cadence, stride length and time, step length and time will be assessed with inertial sensors (OPAL system) for tDCS and SHAM (secondary outcomes). Furthermore, the investigators will calculate the distance walked index (DWI, distance Min 1 - distance Min 6), which is an objective measure of fatigability. A tDCS device (ActivaDose II) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm,soaked with 15 mM NaCL). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit. The following sessions will be performed in randomized order. Group 1 (During) - (A) The participant will receive tDCS or SHAM throughout the walking. In the tDCS trial the intensity will start at 0 mA and will be increased to 2mA over a 30 second period of time. At the 6:30 minute time point (immediately after walking) the current will gradually be reduced from 2 mA to 0 mA. (B) In the sham condition the participants will only receive the initial 30 seconds of stimulation, after which the current will be set to 0. Group 2 (Before) - (C) After a 30s ramp-up, tDCS will be delivered for 13 minutes at an intensity of 2 mA before the 6 min walk test. At the 13:00 minute time point the current will gradually be reduced from 2 mA to 0 mA. (D) Participants who undergo a sham condition will only receive the initial 30 seconds of ramp-up, after which the current will be set to 0 (D). In session 3, the condition not performed during session 2 will be performed. E.g., if a patient in Group 1 was randomly assigned DURING_SHAM for session 2, the patient will perform DURING_tDCS in session 3. All other testing conditions will be the same as session 2.

There will be no long-term follow up.

ELIGIBILITY:
Inclusion Criteria:

* medically diagnosed with Multiple Sclerosis,
* moderate disability (Patient Determined Disease Steps (PDDS) core 2-6), -self-- reported differences in function between legs, able to walk for 6min. -

Exclusion Criteria:

* relapse within last 60 days,
* high risk for cardiovascular disease (ACSM risk classification),
* changes in disease modifying medications within last 45 days,
* concurrent neurological/neuromuscular disease,
* hospitalization within last 90 days,
* diagnosed depression, inability to understand/sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2019-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Rudroff, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Workman CD, Kamholz J, Rudroff T. Transcranial Direct Current Stimulation (tDCS) to Improve Gait in Multiple Sclerosis: A Timing Window Comparison. Front Hum Neurosci. 2019 Nov 28;13:420. doi: 10.3389/fnhum.2019.00420. eCollection 2019. PMID 31849628

RESULTS

PARTICIPANT FLOW:
Groups:
- BEFORE Walking, SHAM First Then tDCS: In the BEFORE walking group, received SHAM in session two and tDCS in session three.
- BEFORE Walking, tDCS First Then SHAM: In the BEFORE walking group, received tDCS in session two and then SHAM in session three.
- DURING Walking, SHAM First Then tDCS: In the DURING walking group, received SHAM in session two and then tDCS in session three.
- DURING Walking, tDCS First Then SHAM: In the DURING walking group, received tDCS in session two and then SHAM in session three.
Period: Overall Study
Arm/Group | BEFORE Walking, SHAM First Then tDCS | BEFORE Walking, tDCS First Then SHAM | DURING Walking, SHAM First Then tDCS | DURING Walking, tDCS First Then SHAM
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Before Walking tDCS/SHAM; During Walking tDCS/SHAM: To investigate the effects of tDCS applied before walking versus during to evaluate effectiveness of the intervention.
  tDCS: Brain Stimulation
  To investigate the effects of SHAM applied before walking versus during to evaluate effectiveness of the intervention.
  SHAM: Placebo device
- Total: Total of all reporting groups
Arm/Group | Before Walking tDCS/SHAM | During Walking tDCS/SHAM | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (14) | 56 (7) | 51 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Distance Walked on a Treadmill With tDCS
Description: 6 min walk test
Time Frame: one week
Measure: Mean (Standard Deviation); unit: m
Groups:
- Before Walking: To investigate the effects of tDCS applied before walking to evaluate effectiveness of the intervention.
  tDCS: Brain Stimulation
  SHAM: Placebo device
- During Walking: To investigate the effects of tDCS applied during to evaluate effectiveness of the intervention.
  tDCS: Brain Stimulation
  SHAM: Placebo device
Arm/Group | Before Walking | During Walking
Number analyzed (Participants) | 6 | 6
m | 375 (78) | 285 (131)

2. Primary Outcome: Distance Walked on a Treadmill With SHAM
Description: 6 min walk test
Time Frame: one week
Measure: Mean (Standard Deviation); unit: m
Groups:
- Before Walking: To investigate the effects of SHAM applied before walking to evaluate effectiveness of the intervention.
  tDCS: Brain Stimulation
  SHAM: Placebo device
- During Walking: To investigate the effects of SHAM applied during walking to evaluate effectiveness of the intervention.
  tDCS: Brain Stimulation
  SHAM: Placebo device
Arm/Group | Before Walking | During Walking
Number analyzed (Participants) | 6 | 6
m | 366 (90) | 298 (133)

3. Other Pre Specified Outcome: Leg Strength Data
Description: Leg extensor strength and Leg flexor strength data were obtained but have not been used for data analysis.
Time Frame: one week
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 weeks.
Groups:
- Before Walking Active/SHAM: To investigate the effects of tDCS applied before walking to evaluate effectiveness of the intervention.
  tDCS: Brain Stimulation
  SHAM: Placebo device
- During Walking Active/SHAM: To investigate the effects of tDCS applied during walking to evaluate effectiveness of the intervention.
  tDCS: Brain Stimulation
  SHAM: Placebo device
Arm/Group | Before Walking Active/SHAM | During Walking Active/SHAM
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT03757819/Prot_SAP_ICF_004.pdf